CLINICAL TRIAL: NCT01123291
Title: Randomized Evaluation of Routine Follow-up Coronary Angiography After Percutaneous Coronary Intervention Trial
Brief Title: Evaluation of Routine Follow-up Coronary Angiography After Percutaneous Coronary Intervention Trial
Acronym: ReACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C406
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: follow-up coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- routine follow-up coronary angiography (Active Comparator): routine follow-up coronary angiography at 8-12 after discharge for percutaneous coronary intervention
  Interventions: Procedure: follow-up coronary angiography
- clinical follow-up (Active Comparator): no routine follow-up coronary angiography at 8-12 after discharge for percutaneous coronary intervention
  Interventions: Procedure: Clinical follow-up

INTERVENTIONS:
Procedure: follow-up coronary angiography — follow-up coronary angiography at 8-12 months after discharge for percutaneous coronary intervention
  Arms: routine follow-up coronary angiography
Procedure: Clinical follow-up — no routine follow-up coronary angiography at 8-12 months after discharge for percutaneous coronary intervention
  Arms: clinical follow-up

SUMMARY:
The purpose of this study is to evaluate the long term clinical impact of routine follow-up coronary angiography after percutaneous coronary intervention (PCI). The primary endpoint is a composite of death/myocardial infarction/stroke/emergency hospitalization for acute coronary syndrome/hospitalization for congestive heart failure at 3-year after percutaneous coronary intervention.

DETAILED DESCRIPTION:
Routine follow-up coronary angiography after percutaneous coronary intervention has been performed to detect restenosis in a lot of PCI centers in Japan. On the other hand, previous studies reported that routine follow-up coronary angiography might lead to unnecessary reinterventions in asymptomatic patients. In this situation, the effect of routine follow-up coronary angiography on long-term clinical outcomes remains unknown. The purpose of this study is to evaluate the long-term clinical impact of routine follow-up coronary angiography after PCI compared with clinical follow-up alone. The primary endpoint of this study is a composite of death/myocardial infarction/stroke/emergency hospitalization for acute coronary syndrome/hospitalization for congestive heart failure at three-year after percutaneous coronary intervention. The design of this study is almost all-comer design enrolling patients received PCI without any exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients received percutaneous coronary intervention
* Patients older than 20 years old
* Patients who will not scheduled any staged percutaneous coronary intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
a composite of death/myocardial infarction/stroke/emergency hospitalization for acute coronary syndrome/hospitalization for congestive heart failure | 4.8 years
  a composite of death/myocardial infarction/stroke/emergency hospitalization for acute coronary syndrome/hospitalization for congestive heart failure

SECONDARY OUTCOMES:
death | 4.8 years
  death
cardiac death | 4.8 years
  cardiac death
myocardial infarction | 4.8 years
  myocardial infarction
stent thrombosis | 4.8 years
  stent thrombosis defined bya Academic Reseach Consortium
stroke | 4.8 years
  both ischemic and hemorrhagic stroke excluding transient ischemic attach
bleeding complications | 4.8 years
  bleeding complications defined by GUSTO and TIMI
any coronary revascularization | 4.8 years
  any coronary revascularization
clinically-driven coronary revascularization | 4.8 years
  clinically-driven coronary revascularization
clinically-driven target-lesion revascularization | 4.8 years
  clinically-driven target-lesion revascularization
any target-lesion revascularization | 4.8 years
  any target-lesion revascularization
coronary artery bypass grafting | 4.8 years
  coronary artery bypass grafting
angina | 4.8 years
  angina
renal function | 4.8 years
  estimate-glomerular filtration rate
emergency hospitalization for acute coronary syndrome | 4.8 years
  emergency hospitalization for acute coronary syndrome
hospitalization for congestive heart failure | 4.8 years
  hospitalization for congestive heart failure
composite of cardiac death, myocardial infarction or acute coronary syndrome | 4.8 years
  composite of cardiac death, myocardial infarction or acute coronary syndrome
follow-up coronary angiography | 4.8 years
  presence of follow-up coronary angiography
clinically-driven follow-up coronary angiography | 4.8 years
  presence of clinically-driven follow-up coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, Principal Investigator — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Division of Cardiology, Kyoto University Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Shiomi H, Morimoto T, Kitaguchi S, Nakagawa Y, Ishii K, Haruna Y, Takamisawa I, Motooka M, Nakao K, Matsuda S, Mimoto S, Aoyama Y, Takeda T, Murata K, Akao M, Inada T, Eizawa H, Hyakuna E, Awano K, Shirotani M, Furukawa Y, Kadota K, Miyauchi K, Tanaka M, Noguchi Y, Nakamura S, Yasuda S, Miyazaki S, Daida H, Kimura K, Ikari Y, Hirayama H, Sumiyoshi T, Kimura T; ReACT Investigators. The ReACT Trial: Randomized Evaluation of Routine Follow-up Coronary Angiography After Percutaneous Coronary Intervention Trial. JACC Cardiovasc Interv. 2017 Jan 23;10(2):109-117. doi: 10.1016/j.jcin.2016.10.018. Epub 2016 Dec 28. PMID 28040445